CLINICAL TRIAL: NCT04306354
Title: Randomized, Double-Blind, Placebo Controlled Study of Intranasal Oxytocin During Detoxification of Crack Cocaine
Brief Title: Use of Intranasal Oxytocin During Detoxification of Crack Cocaine
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontificia Universidade Católica do Rio Grande do Sul (Other)
Collaborators: Secretaria Nacional de Políticas sobre Drogas (SENAD) (Unknown); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Rodrigo Grassi-Oliveira, Professor, Pontificia Universidade Católica do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U1111-1188-6555; U1111-1188-6555 (Registry Identifier: Registro Brasileiro de Ensaios Clínicos); 39868314.0.0000.5336 (Registry Identifier: Plataforma Brasil)
Record Dates: First submitted 2020-03-09; First posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Cocaine Withdrawal; Cocaine Smoking; Cocaine-Related Disorders
Keywords: crack cocaine; addiction; stimulants; oxytocin; detoxification; abstinence; withdrawal
MeSH Terms: conditions — Cocaine Smoking; Cocaine-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: On the eve of the eighth day of hospitalization, a person in charge of the research team performed a randomization of the participants exchanged in blocks, according to the methods of Schulz and collaborators (SCHULZ; GRIMES, 2002). The responsible person did not have contact with the participants. The blocks were made up of 12 participants each, and the ratio was maintained at 4: 4: 4, in order to reduce the chances of the groups getting mixed amounts. The members of the research team responsible for data collection, the technical team of the inpatient unit and the participants did not know to what condition each patient had been allocated.
  These procedures guaranteed the randomization and double blinding of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Conventional oxytocin treatment (T + OC) (Experimental): 32 female cocaine users hospitalized for detoxification will receive six 4 IU jets of intranasal oxytocin twice daily (daily dose of 48 IU) as adjunctive treatment to conventional treatment from the eighth to seventeenth day of hospitalization (duration of oxytocin treatment of 10 days). Conventional treatment includes supportive individual and group psychotherapy (once a week), nutritional control, regular physical activity and psychopharmacotherapy as needed to relieve the symptoms of anxiety, aggression and agitation typical of withdrawal and care. 21 days of hospitalization.
  Interventions: Drug: Oxytocin nasal spray
- Conventional treatment with placebo administration (T + PBO) (Placebo Comparator): 32 female cocaine users hospitalized for detoxification will receive six jets of placebo solution (2% odor-generating propolis essence + the same vehicle as intra-nasal oxytocin: 0.05% citric acid, 0.9% sodium chloride, 1% glycerol, 0.54% disodium phosphate, 0.2% methylparaben + propylparaben, 1% sorbitol, 80% water) twice daily as adjunctive treatment to conventional treatment from the eighth to the seventeenth day of hospitalization (duration of placebo treatment of 10 days). Conventional treatment includes supportive individual and group psychotherapy (once a week), nutritional control, regular physical activity and psychopharmacotherapy as needed to relieve the symptoms of anxiety, aggression and agitation typical of withdrawal and care. 21 days of hospitalization.
  Interventions: Drug: placebo nasal spray
- Conventional treatment (T) (No Intervention): 32 female cocaine users hospitalized for detoxification will receive conventional treatment including individual and group supportive psychotherapy (once a week), nutritional control, regular physical activity and psychopharmacotherapy if needed for symptom relief. anxiety, aggression and agitation, typical of abstinence and nursing care, during 21 days of hospitalization.

INTERVENTIONS:
Drug: Oxytocin nasal spray — Oxytocin nasal spray 24 UI twice daily as adjunctive treatment to conventional treatment during 10 days of detoxification of crack cocaine
  Arms: Conventional oxytocin treatment (T + OC)
Drug: placebo nasal spray — Nasal spray with placebo solution (2% odor-generating propolis essence + the same vehicle as intra-nasal oxytocin: 0.05% citric acid, 0.9% sodium chloride, 1% glycerol, 0.54% disodium phosphate, 0.2% methylparaben + propylparaben, 1% sorbitol, 80% water) twice daily as adjunctive treatment to conventional treatment.
  Arms: Conventional treatment with placebo administration (T + PBO)

SUMMARY:
Randomized treatment control trial, double-blind, parallel, with two arms including ninety-six hospitalized women between 18 and 52 years. Those who agree to participate in the study and meet the eligibility criteria will be randomly allocated to one of the following experimental conditions:

* Conventional oxytocin treatment (T + OC): 32 female cocaine users hospitalized for detoxification will receive six 4 IU jets of intranasal oxytocin twice daily (daily dose of 48 IU) as adjunctive treatment to conventional treatment from the eighth to seventeenth day of hospitalization (duration of oxytocin treatment of 10 days). Conventional treatment includes supportive individual and group psychotherapy (once a week), nutritional control, regular physical activity and psychopharmacotherapy as needed to relieve the symptoms of anxiety, aggression and agitation typical of withdrawal and care. 21 days of hospitalization.
* Conventional treatment with placebo administration (T + PBO): 32 female cocaine users hospitalized for detoxification will receive six jets of placebo solution (2% odor-generating propolis essence + the same vehicle as intra-nasal oxytocin: 0.05% citric acid, 0.9% sodium chloride, 1% glycerol, 0.54% disodium phosphate, 0.2% methylparaben + propylparaben, 1% sorbitol, 80% water) twice daily as adjunctive treatment to conventional treatment from the eighth to the seventeenth day of hospitalization (duration of placebo treatment of 10 days). Conventional treatment includes supportive individual and group psychotherapy (once a week), nutritional control, regular physical activity and psychopharmacotherapy as needed to relieve the symptoms of anxiety, aggression and agitation typical of withdrawal and care. 21 days of hospitalization.
* Conventional treatment (T): 32 female cocaine users hospitalized for detoxification will receive conventional treatment including individual and group supportive psychotherapy (once a week), nutritional control, regular physical activity and psychopharmacotherapy if needed for symptom relief. anxiety, aggression and agitation, typical of abstinence and nursing care, during 21 days of hospitalization.

Outcomes: Withdrawal symptoms, Anxiety symptoms and Depressive symptoms

DETAILED DESCRIPTION:
Design: Randomized treatment control trial, double-blind, parallel, with two arms.

Sample: Ninety-six hospitalized women between 18 and 52 years will participate in this study. Those who agree to participate in the study and meet the eligibility criteria will be randomly allocated to one of the following experimental conditions:

* Conventional oxytocin treatment (T + OC): 32 female cocaine users hospitalized for detoxification will receive six 4 IU jets of intranasal oxytocin twice daily (daily dose of 48 IU) as adjunctive treatment to conventional treatment from the eighth to seventeenth day of hospitalization (duration of oxytocin treatment of 10 days). Conventional treatment includes supportive individual and group psychotherapy (once a week), nutritional control, regular physical activity and psychopharmacotherapy as needed to relieve the symptoms of anxiety, aggression and agitation typical of withdrawal and care. 21 days of hospitalization.
* Conventional treatment with placebo administration (T + PBO): 32 female cocaine users hospitalized for detoxification will receive six jets of placebo solution (2% odor-generating propolis essence + the same vehicle as intra-nasal oxytocin: 0.05% citric acid, 0.9% sodium chloride, 1% glycerol, 0.54% disodium phosphate, 0.2% methylparaben + propylparaben, 1% sorbitol, 80% water) twice daily as adjunctive treatment to conventional treatment from the eighth to the seventeenth day of hospitalization (duration of placebo treatment of 10 days). Conventional treatment includes supportive individual and group psychotherapy (once a week), nutritional control, regular physical activity and psychopharmacotherapy as needed to relieve the symptoms of anxiety, aggression and agitation typical of withdrawal and care. 21 days of hospitalization.
* Conventional treatment (T): 32 female cocaine users hospitalized for detoxification will receive conventional treatment including individual and group supportive psychotherapy (once a week), nutritional control, regular physical activity and psychopharmacotherapy if needed for symptom relief. anxiety, aggression and agitation, typical of abstinence and nursing care, during 21 days of hospitalization.

Inclusion Criteria:

* Volunteers (no payment to be enroll in the research according with Brazilian legislation)
* Age 18-52 years
* Primary diagnosis of cocaine crack dependence according to DSM-5
* Sex feminine
* Participants must be abstinent at least 7 days prior the study intervention
* Participants must consent to be randomly allocated to experimental conditions

Exclusion Criteria:

* Pregnancy
* Puerperium
* Breastfeeding
* Menopause
* Currently using hormone therapy
* Total hysterectomy
* Diagnosis or suspicion of autoimmune or neurological diseases and / or syndromes (stroke, Parkinson and Alzheimer's)
* Diagnosis or suspected current decompensated and / or severe endocrine, cardiovascular, pulmonary, renal, gastrointestinal disorders
* Moderate or severe psychotic syndrome
* Obesity Level III
* Intellectual impairment (IQ <70)
* Corticosteroid therapy, glucocorticoid or any exogenous steroid therapy
* Infectious condition or acute febrile syndrome
* Significant nasal congestion
* Type III nasal septum deviation (cases considered severe with deviated septum in which breathing is impaired)
* Mucosal lesions
* History of head trauma moderate or severe (Glasgow <12)
* HIV +

Primary Outcome Measure:

1. Withdrawal symptoms Change from baseline withdrawal symptoms (hospital admission) at the end of detoxification treatment (21 days) assessed by Cocaine Selective Severity Assessment (CSSA, minimum and maximum scores: 0 - 112). After treatment, the oxytocin-treated group is expected to have significantly lower withdrawal scores (better outcome) than the other groups (30%).
2. Anxiety symptoms Change from baseline anxiety symptoms (hospital admission) at the end of detoxification treatment (21 days) assessed by the Patient-Reported Outcomes Measurement Information System Short Form scale (PROMIS, minimum and maximum raw scores: 8 - 40). After treatment, the oxytocin-treated group is expected to show lower anxiety scores (better outcome) compared to the other groups (30%).
3. Depression symptoms Change from baseline depressive symptoms (hospital admission) at the end of detoxification treatment (21 days) assessed by the Quick Inventory of Depressive Symptomatology Self-Report scale (QIDS-SR, minimum and maximum scores: 0 - 27). After treatment, the oxytocin-treated group is expected to show lower depressive scores (better outcome) compared to the other groups (30%).

Secondary Outcome Measures:

1. Neuroleptic Dose Change Dose change of neuroleptic medications used during hospitalization for agitation or irritability (expected 25% lower).
2. Adherence of outpatient treatment Rate of adherence of outpatient treatment six months after discharge (expected to be 20% higher) assessed by reviewing the medical records of each patient within the outpatient program. If patient would be enrolled in the outpatient program after six months from detoxification she will be considered adhered to the program (higher rates means better outcome).

ELIGIBILITY:
Inclusion Criteria:

* Volunteers (no payment to be enroll in the research according with Brazilian legislation)
* Age 18-52 years
* Primary diagnosis of cocaine crack dependence according to DSM-5
* Sex feminine
* Participants must be abstinent at least 7 days prior the study intervention
* Participants must consent to be randomly allocated to experimental conditions

Exclusion Criteria:

* Pregnancy
* Puerperium
* Breastfeeding
* Menopause
* Currently using hormone therapy
* Total hysterectomy
* Diagnosis or suspicion of autoimmune or neurological diseases and / or syndromes (stroke, Parkinson and Alzheimer's)
* Diagnosis or suspected current decompensated and / or severe endocrine, cardiovascular, pulmonary, renal, gastrointestinal disorders
* Moderate or severe psychotic syndrome
* Obesity Level III
* Intellectual impairment (IQ <70)
* Corticosteroid therapy, glucocorticoid or any exogenous steroid therapy
* Infectious condition or acute febrile syndrome
* Significant nasal congestion
* Type III nasal septum deviation (cases considered severe with deviated septum in which breathing is impaired)
* Mucosal lesions
* History of head trauma moderate or severe (Glasgow <12)
* HIV +

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2018-09-15 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Withdrawal symptoms | Change from baseline (first week after hospital admission) at the end of detoxification treatment (21 days).
  Change from baseline withdrawal symptoms (hospital admission) at the end of detoxification treatment (21 days) assessed by Cocaine Selective Severity Assessment (CSSA, minimum and maximum scores: 0 - 112). After treatment, the oxytocin-treated group is expected to have significantly lower withdrawal scores (better outcome) than the other groups (30%).
Anxiety symptoms | Change from baseline (first week after hospital admission) at the end of detoxification treatment (21 days).
  Change from baseline anxiety symptoms (hospital admission) at the end of detoxification treatment (21 days) assessed by the Patient-Reported Outcomes Measurement Information System Short Form scale (PROMIS, minimum and maximum raw scores: 8 - 40). After treatment, the oxytocin-treated group is expected to show lower anxiety scores (better outcome) compared to the other groups (30%).
Depression symptoms | Change from baseline (first week after hospital admission) at the end of detoxification treatment (21 days).
  Change from baseline depressive symptoms (hospital admission) at the end of detoxification treatment (21 days) assessed by the Quick Inventory of Depressive Symptomatology Self-Report scale (QIDS-SR, minimum and maximum scores: 0 - 27). After treatment, the oxytocin-treated group is expected to show lower depressive scores (better outcome) compared to the other groups (30%).

SECONDARY OUTCOMES:
Neuroleptic Dose Change | Change from baseline (first week after hospital admission) at the end of detoxification treatment (21 days)
  Dose change of neuroleptic medications used during hospitalization for agitation or irritability (expected 25% lower).
Adherence of outpatient treatment | six months after hospital discharge
  Rate of adherence of outpatient treatment six months after discharge (expected to be 20% higher) assessed by reviewing the medical records of each patient within the outpatient program. If patient would be enrolled in the outpatient program after six months from detoxification she will be considered adhered to the program (higher rates means better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Grassi-Oliveira, MD, PhD, Principal Investigator — Pontifícia Universidade Católica do Rio Grande do Sul
Locations (1):
- Hospital Santa Ana, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: By the time of publication
Access Criteria: open access